CLINICAL TRIAL: NCT02243540
Title: Impact of Bladder Underactivity on Treatment Outcomes of Laser Prostatectomy: Comparison Between Potassium-titanyl-phosphate Photoselective Vaporization of the Prostate (PVP) and Holmium Laser Enucleation of the Prostate (HoLEP)
Brief Title: Impact of Bladder Underactivity on Treatment Outcomes of Laser Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Seung Paick, Professor, Seoul National University Hospital
Other Study IDs: JSPaick1
Record Dates: First submitted 2014-09-14; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to evaluate an impact of preoperative bladder underactivity on treatment outcomes of photoselective vaporization of the prostate (PVP) or holmium laser enucleation of the prostate (HoLEP) in the treatment of benign prostatic obstruction, and to compare it between the two types of surgery for benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* patients in whom 12-month follow-up data were available

Exclusion Criteria:

* a previous diagnosis of urethral stricture
* prostate or bladder carcinoma
* neurogenic bladder disease
* a previous history of urological surgery

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men who underwent photoselective vaporization of the prostate (PVP) or holmium laser enucleation of the prostate (HoLEP) for benign prostatic hyperplasia refractory to medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 1828 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline bladder voiding efficiency at 12 months after surgery | 12-months postoperatively
  bladder voiding efficiency = voided volume x 100 / (voided volume + post-void residual urine volume)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Seung Paick, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea